CLINICAL TRIAL: NCT04264728
Title: Adult-onset Generalized Morphea : A Retrospective Multicenter Study
Brief Title: Adult-onset Generalized Morphea
Acronym: MORPHEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7551
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Generalized Morphea
Keywords: Morphea; Generalized Morphea; Localized Scleroderma
MeSH Terms: conditions — Scleroderma, Localized

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to describe the demographical and clinical characteristics of a retrospective cohort of adult-onset GM and to investigate whether these findings differ between patients with an isomorphic and a symmetric pattern of lesion distribution.

ELIGIBILITY:
Inclusion Criteria:

* Age of onset ≥ 18 years
* Patients with generalized morphea as defined by criteria established by Laxer and Zulian (4 or more morpheaform plaques larger than 3 centimeters that show tendency to confluence and involve at least 2 different anatomic sites)
* Availability of good-quality clinical photographs
* Patient who, after being informed, has not expressed his or her opposition to the re-use of his or her data for the purposes of this research

Exclusion Criteria:

* Patients with linear morphea who met criteria for generalized morphea
* Patient's opposition to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient with generalized morphea as defined by criteria established by Laxer and Zulian (4 or more morpheaform plaques larger than 3 centimeters that show tendency to confluence and involve at least 2 different anatomic sites)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of generalized morphea in adult patients consulted in dermatology departments | Files analyzed retrospectily from January 1st, 2019 to September 30, 2019 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Cédric LENORMAND, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de dermatologie - Hôpital Civil de Strasbourg, Strasbourg, France